CLINICAL TRIAL: NCT03260543
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Fermented Ginseng Powder on Liver Function
Brief Title: Efficacy and Safety of Fermented Ginseng Powder on Liver Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GB-LFE-GP
Record Dates: First submitted 2017-03-23; First posted 2017-08-24 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Fatty Liver, Nonalcoholic
Keywords: ginseng powder; Fatty Liver; Clinical Trial
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fermented ginseng powder (Experimental): tablets (2 tablets/day, 125 mg & 500 mg/day) for 12 weeks.
  Interventions: Dietary Supplement: fermented ginseng powder
- Placebo (Placebo Comparator): Placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fermented ginseng powder — tablets (2 tablets/day, 125 mg & 500 mg/day) for 12 weeks.
  Arms: fermented ginseng powder
Dietary Supplement: Placebo — Placebo for 12 weeks.
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of fermented ginseng powder on improvement of Liver function.

DETAILED DESCRIPTION:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of fermented ginseng powder on improvement of Liver function. The investigators measured ALT(Alanine Transaminase) profiles, Liver function index, fatty liver grade, lipid metabolism index, total antioxidant capacity, imflammation index, and Multidimensional Fatigue Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-70 years with ALT 35-105 IU/L

Exclusion Criteria:

* Under antipsychotic drugs therapy within past 2 months
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test by show the following results

  * Serum Creatinine > 2.0 mg/dl
* Pregnancy or breast feeding etc.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes of ALT(Alanine Transaminase) | Baseline and 12 weeks
  Changes of ALT were assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of Liver function index | Baseline and 12 weeks
  Changes of AST were assessed before and after the intervention
Changes of fatty liver grade | Baseline and 12 weeks
  Changes of fatty liver grade were assessed before and after the intervention
Changes of lipid metabolism index | Baseline and 12 weeks
  Changes of lipid metabolism index were assessed before and after the intervention
Changes of total antioxidant capacity | Baseline and 12 weeks
  Changes of total antioxidant capacity were assessed before and after the intervention
Changes of imflammation index | Baseline and 12 weeks
  Changes of imflammation index were assessed before and after the intervention
Changes of Multidimensional Fatigue Scale | Baseline and 12 weeks
  Changes of Multidimensional Fatigue Scale were assessed before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jung SJ, Hwang JH, Park SH, Choi EK, Ha KC, Baek HI, Shin DG, Seo JH, Chae SW. A 12-week, randomized, double-blind study to evaluate the efficacy and safety of liver function after using fermented ginseng powder (GBCK25). Food Nutr Res. 2020 Apr 6;64. doi: 10.29219/fnr.v64.3517. eCollection 2020. PMID 32425736